CLINICAL TRIAL: NCT04814459
Title: Prevention Focused Home-Based Physical Therapy Utilizing Community Partnership Referrals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oakland University (Other)
Collaborators: Michigan Health Endowment Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 912215-18
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Results first posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-09

CONDITIONS: Fall; Risk Reduction
Keywords: Older adults
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Intervention Model Description: Experimental group (EG) participated in the 7-month HOP-UP-PT control group (CG) included only baseline, 3-month, and 7-month assessments. The CG was instructed to continue their normal level of activity throughout the 7-months after which they were offered the opportunity to receive the HOP-UP-PT program. This study reports only the 7-month time frame during which the EG and CG can be directly compared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOP-UP-PT Program (Experimental): HOP-UP-PT Program group will participate in the 7-month HOP-UP-PT program
  Interventions: Other: HOP-UP-PT Program
- Normal Level of Activity (No Intervention): Normal Level of Activity group will be instructed to continue their normal level of activity throughout the 7-months after which they will be offered the opportunity to receive the HOP-UP-PT program

INTERVENTIONS:
Other: HOP-UP-PT Program — Interventions provided to EG participants included; (1) the Otago Exercise Program (OEP) which is a well-established exercise program with evidence that it reduces falls among community-dwelling older adults, (2) motivational interviewing (MI) to optimize positive health behaviors, and (3) home and environmental modification recommendations aimed at safety. Participants were provided with and educated on the use of a wrist-worn activity tracker and an automated BP monitor unit. Finally, when follow up items were identified (e.g., orthostatic hypotension, community exercise classes), these referrals were made and documented.
  Arms: HOP-UP-PT Program

SUMMARY:
This novel study supports the positive benefits of Home Based Older Persons Upstreaming Physical Therapy (HOP-UP-PT) to older adults identified as "at-risk" by their local senior center after participating in a prevention-focused multimodal program provided by physical therapists in their home.

DETAILED DESCRIPTION:
The purpose of this study was to describe the outcomes of Home Based Older Persons Upstreaming Physical Therapy (HOP-UP-PT) program participants and then to compare these outcomes to non-participants. 144 participants (n=72 per group) will be randomized to either the HOP-UP-PT intervention group or the Normal level of activity group. Six Michigan senior centers will refer adults ≥ 65 years who were at-risk for functional decline or falls. Licensed physical therapists will deliver physical, environmental, and health interventions within their approved scope of practice to the HOP-UP-PT intervention group during nine encounters (six in-person, three telerehabilitation) delivered over seven months. The Normal level of activity group participants are told to continue their usual physical activity routines during the same timeframe. Baseline and re-assessments are conducted at 0-, 3-, and 7-months for both the HOP-UP-PT intervention group and Normal level of activity group. Descriptions and comparisons from each assessment encounter will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 65 years of age
* Senior Community Center staff identified them as 'at-risk' for decline in community dwelling status due to physical, social, economic, or community-related barriers
* Willingness to participate

Exclusion Criteria:

* Received physical therapy services within the prior two months in any setting
* Had been hospitalized within the prior two months
* Were currently receiving palliative or hospice care
* Mini Cog score less than 4 and Trail Making Part B score greater than 273 seconds
* Outcomes American College of Sports Medicine exercise pre-participation health screening indicating physician clearance needed for participation and after evaluation the physician will not clear

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Arena, DScPT, Principal Investigator — Oakland University
Locations (1):
- Oakland University, Rochester, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared

REFERENCES:
- [Background] Wilson CM, Arena SK, Adcock K, Colling D. A Home-Based Older Person Upstreaming Prevention Physical Therapy (HOP-UP-PT) Program Utilizing Community Partnership Referrals. Home Healthc Now. 2019 Mar/Apr;37(2):88-96. doi: 10.1097/NHH.0000000000000716. PMID 30829786
- [Background] Arena SK, Wilson CM, Peterson E. Targeted Population Health Utilizing Direct Referral to Home-Based Older Person Upstreaming Prevention Physical Therapy From a Community-Based Senior Center. Cardiopulm Phys Ther J. 2020;31(1):11-21. doi:10.1097/CPT.0000000000000131
- [Background] Wilson C, Arena SK, Starceski R, Swanson K. Older Adults' Outcomes and Perceptions After Participating in the HOP-UP-PT Program: A Prospective Descriptive Study. Home Healthc Now. 2020 Mar/Apr;38(2):86-91. doi: 10.1097/NHH.0000000000000843. PMID 32134816
- [Background] Measuring orthostatic blood pressure. Center for Disease Control and Prevention. Published 2017. https://www.cdc.gov/steadi/materials.html
- [Background] Hill KD, Schwarz JA, Kalogeropoulos AJ, Gibson SJ. Fear of falling revisited. Arch Phys Med Rehabil. 1996 Oct;77(10):1025-9. doi: 10.1016/s0003-9993(96)90063-5. PMID 8857881
- [Background] Black B, Marcoux BC, Stiller C, Qu X, Gellish R. Personal health behaviors and role-modeling attitudes of physical therapists and physical therapist students: a cross-sectional study. Phys Ther. 2012 Nov;92(11):1419-36. doi: 10.2522/ptj.20110037. Epub 2012 Jul 19. PMID 22822236
- [Background] Groll DL, To T, Bombardier C, Wright JG. The development of a comorbidity index with physical function as the outcome. J Clin Epidemiol. 2005 Jun;58(6):595-602. doi: 10.1016/j.jclinepi.2004.10.018. PMID 15878473
- [Background] Adult BMI Calculator. Center for Disease Control and Prevention. Published 2020. Accessed January 25, 2021. https://www.cdc.gov/healthyweight/assessing/bmi/adult_bmi/english_bmi_calculator/bmi_calculator.html
- [Background] STEADI: Algorithm for FallRisk Screening, Assessment, and Intervention. Center for Disease Control and Prevention. Published 2017. Accessed January 28, 2019. https://www.cdc.gov/steadi/materials.html
- [Background] Mackenzie L, Byles J, Higginbotham N. Reliability of the Home Falls and Accidents Screening Tool (HOME FAST) for identifying older people at increased risk of falls. Disabil Rehabil. 2002 Mar 20;24(5):266-74. doi: 10.1080/09638280110087089. PMID 12004972
- [Background] Shumway-Cook A, Baldwin M, Polissar NL, Gruber W. Predicting the probability for falls in community-dwelling older adults. Phys Ther. 1997 Aug;77(8):812-9. doi: 10.1093/ptj/77.8.812. PMID 9256869
- [Background] Four Stage Balance Test. Center for Disease Control and Prevention. Published 2017. Accessed January 25, 2021. https://www.cdc.gov/steadi/pdf/4-Stage_Balance_Test-print.pdf
- [Background] Macfarlane DJ, Chou KL, Cheng YH, Chi I. Validity and normative data for thirty-second chair stand test in elderly community-dwelling Hong Kong Chinese. Am J Hum Biol. 2006 May-Jun;18(3):418-21. doi: 10.1002/ajhb.20503. PMID 16634026
- [Background] Five Time Sit to Stand Test. Shirley Ryan Ability Lab. Published 2021. Accessed January 25, 2021. https://www.sralab.org/rehabilitation-measures/five-times-sit-stand-test
- [Background] Tiedemann A, Shimada H, Sherrington C, Murray S, Lord S. The comparative ability of eight functional mobility tests for predicting falls in community-dwelling older people. Age Ageing. 2008 Jul;37(4):430-5. doi: 10.1093/ageing/afn100. Epub 2008 May 16. PMID 18487264
- [Background] Pavasini R, Guralnik J, Brown JC, di Bari M, Cesari M, Landi F, Vaes B, Legrand D, Verghese J, Wang C, Stenholm S, Ferrucci L, Lai JC, Bartes AA, Espaulella J, Ferrer M, Lim JY, Ensrud KE, Cawthon P, Turusheva A, Frolova E, Rolland Y, Lauwers V, Corsonello A, Kirk GD, Ferrari R, Volpato S, Campo G. Short Physical Performance Battery and all-cause mortality: systematic review and meta-analysis. BMC Med. 2016 Dec 22;14(1):215. doi: 10.1186/s12916-016-0763-7. PMID 28003033
- [Background] Fritz S, Lusardi M. White paper: "walking speed: the sixth vital sign". J Geriatr Phys Ther. 2009;32(2):46-9. No abstract available. PMID 20039582
- [Background] Campbell A RM. Otago Exercise Program to Prevent Falls in Older Adults. Otago Medical School, University of Otago. Accessed January 25, 2021. https://www.livestronger.org.nz/assets/Uploads/acc1162-otago-exercise-manual.pdf
- [Background] Kyrdalen IL, Moen K, Roysland AS, Helbostad JL. The Otago Exercise Program performed as group training versus home training in fall-prone older people: a randomized controlled Trial. Physiother Res Int. 2014 Jun;19(2):108-16. doi: 10.1002/pri.1571. Epub 2013 Dec 11. PMID 24339273
- [Background] Pignataro RM, Huddleston J. The Use of Motivational Interviewing in Physical Therapy Education and Practice: Empowering Patients Through Effective Self-Management. J Phys Ther Educ. 2015;29(2):62-71. doi:10.1097/00001416-201529020-00009
- [Derived] Arena SK, Wilson CM, Boright L, Peterson E. Impact of the HOP-UP-PT program on older adults at risk to fall: a randomized controlled trial. BMC Geriatr. 2021 Oct 1;21(1):520. doi: 10.1186/s12877-021-02450-0. PMID 34598692

RESULTS

PARTICIPANT FLOW:
Groups:
- HOP-UP-PT Program: HOP-UP-PT Program group will participate in the 7-month HOP-UP-PT program
  HOP-UP-PT Program: Interventions provided to HOP-UP-PT program participants included; (1) the Otago Exercise Program (OEP) which is a well-established exercise program with evidence that it reduces falls among community-dwelling older adults, (2) motivational interviewing (MI) to optimize positive health behaviors, and (3) home and environmental modification recommendations aimed at safety. Participants were provided with and educated on the use of a wrist-worn activity tracker and an automated BP monitor unit. Finally, when follow up items were identified (e.g., orthostatic hypotension, community exercise classes), these referrals were made and documented.
Period: Overall Study
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Started | 72 | 72
Completed | 72 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HOP-UP-PT Program | Normal Level of Activity | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 72 | 72 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.6 (7.0) | 77.2 (8.2) | 76.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 53 | 110
  Male | 15 | 19 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72 | 72 | 144

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reported Falls
Description: Record of falls in prior year, and between each subsequent visit.
Time Frame: 7 months
Population: Inclusive of low, moderate, and high STEADI fall risk
Measure: Count of Participants; unit: Participants
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Number analyzed (Participants) | 72 | 72
Participants
  Baseline (All Participants) | 37 | 34
  Baseline (Moderat and High STEADI Risk): number analyzed (Participants) | 43 | 39
  Baseline (Moderat and High STEADI Risk) | 29 | 24
  3 Month (All Participants): number analyzed (Participants) | 64 | 60
  3 Month (All Participants) | 5 | 3
  3 Month (Moderate and Hight STEADI Risk): number analyzed (Participants) | 29 | 32
  3 Month (Moderate and Hight STEADI Risk) | 5 | 2
  7 months (All Participants): number analyzed (Participants) | 54 | 56
  7 months (All Participants) | 7 | 15
  7 Month (Moderate and High STEADI Risk): number analyzed (Participants) | 16 | 23
  7 Month (Moderate and High STEADI Risk) | 1 | 11

2. Primary Outcome: Modified Short Physical Performance Battery (SPPB)
Description: The Modified SPPB uses a 0-12 scale (0 = lowest function, 12 = highest function), calculated using collective outcomes of The Four Test Balance Scale (0= unable to perform, 1 = able to stand: feet together >10 sec, 2 = semi-tandem >10 sec, 4 = tandem stance >10 sec, higher score is better balance), 5 Time Sit to Stand (0 = >60 sec, 1=16.7 to 60 sec, 2 = 13.7 to 16.69 sec, 3 = 11.2 to 13.69 sec, and 4 = <11.19 sec, faster time is higher function), and the 3-meter gait speed test (0 = unable to perform, 1= > 6.52 sec, 2 = 4.66 to 6.52 sec, 3 = 3.62 to 4.65 sec, and 4 = < 3.62 sec, faster time is higher function). Each of the three categories has a highest score of 4 and are summed together for a highest total Modified SPPB score of 12.
Time Frame: 7 Months
Population: Data collectors did not complete all measures to calculate this score at the baseline assessment due to variations in patient care delivery. Additionally, participants that were dis-enrolled reduced the data for analysis at the 3 and 7 month encounters.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Number analyzed (Participants) | 72 | 72
score on a scale
  Baseline (all participants): number analyzed (Participants) | 71 | 71
  Baseline (all participants) | 8.44 (2.66) | 7.34 (2.85)
  Baseline (Moderate and high STEADI Risk): number analyzed (Participants) | 42 | 39
  Baseline (Moderate and high STEADI Risk) | 7.64 (2.82) | 6.18 (2.86)
  3 Month (all participants): number analyzed (Participants) | 65 | 53
  3 Month (all participants) | 9.29 (2.49) | 8.04 (2.97)
  3 Month (Moderate and High STEADI Risk): number analyzed (Participants) | 29 | 30
  3 Month (Moderate and High STEADI Risk) | 8.24 (2.43) | 6.60 (2.95)
  7 Month (all participants): number analyzed (Participants) | 48 | 45
  7 Month (all participants) | 9.50 (2.22) | 8.96 (2.63)
  7 Month (Moderate and High STEADI Risk): number analyzed (Participants) | 14 | 20
  7 Month (Moderate and High STEADI Risk) | 7.64 (2.17) | 7.25 (2.67)

3. Primary Outcome: Timed Up and Go
Description: The Timed Up and Go (TUG) is a times assessment of sit to stand transfer, 20 foot bought of ambulation with a 180 degree turn at 10 feet concluding with a stand to sit transfer.
Time Frame: 7 Months
Population: Participants that were dis-enrolled reduced the data available for analysis at the 3 and 7 month encounters.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Number analyzed (Participants) | 72 | 72
seconds
  Baseline (All participants) | 11.5 (4.6) | 13.3 (6.0)
  Baseline (Moderate and High STEADI Risk): number analyzed (Participants) | 42 | 38
  Baseline (Moderate and High STEADI Risk) | 12.9 (5.3) | 15.7 (6.8)
  3 Month (All participants): number analyzed (Participants) | 65 | 57
  3 Month (All participants) | 10.7 (3.7) | 13.0 (6.3)
  3 Month (Moderate and High STEADI Risk): number analyzed (Participants) | 29 | 31
  3 Month (Moderate and High STEADI Risk) | 12.0 (4.3) | 15.4 (7.5)
  7 Month (All participants): number analyzed (Participants) | 54 | 50
  7 Month (All participants) | 10.6 (3.7) | 11.9 (5.4)
  7 Month (Moderate and High STEADI Risk): number analyzed (Participants) | 15 | 22
  7 Month (Moderate and High STEADI Risk) | 13.8 (4.3) | 14.6 (6.8)

4. Primary Outcome: Stopping Elderly Accidents, Death & Injuries (STEADI) Fall Risk Categorization
Description: Low, moderate, and high risk was determined relative to results of the stay independent brochure, subjective report of falls and fall risk and brochure questions, as well as gait, strength, and balance assessment. The Stopping Elderly Accidents, Death & Injuries (STEADI) Algorithm underwent revisions since the study onset, the 2015 version was utilized as a guide for key outcome metrics reported in this study. Low STEADI risk =0, moderate STEADI risk =1, and high STEADI risk = 2. Low risk participants were categorized based on "no" responses to falls or fall risk questions as well as no gait, strength, or balance problems. Moderate risk participants were categorized by answering "yes" to key questions as well as demonstrating some gait, strength, or balance problems, and had a fall without injury. High risk participants were categorized by answering yes to key questions, demonstrating gait, strength, or balance problems, and had 2 or more falls or 1 fall with an injury.
Time Frame: 7 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Number analyzed (Participants) | 72 | 72
score on a scale
  Baseline (All participants): number analyzed (Participants) | 70 | 69
  Baseline (All participants) | 0.8 (0.7) | 0.7 (0.7)
  3 Month (All participants): number analyzed (Participants) | 62 | 54
  3 Month (All participants) | 0.6 (0.7) | 0.7 (0.6)
  7 Month (All Participants): number analyzed (Participants) | 51 | 50
  7 Month (All Participants) | 0.4 (0.6) | 0.6 (0.7)

5. Secondary Outcome: Stay Independent Questionnaire
Description: This questionnaire scores a fall risk on a scale from zero to 14, with 4 or more indicating a possible fall risk. Zero is the lowest fall risk score, 14 is a highest fall risk score.
Time Frame: 3 Months
Population: There is missing data at baseline and 7 month assessment due to data collectors not completing all tests due to variation in patient care performance. Additionally, participants that were dis-enrolled reduced the data available for analysis at the 3 and 7 month encounters.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Number analyzed (Participants) | 72 | 72
score on a scale
  Baseline (All participants): number analyzed (Participants) | 72 | 69
  Baseline (All participants) | 4.8 (3.0) | 4.7 (3.2)
  Baseline (Moderate and High STEADI Risk): number analyzed (Participants) | 43 | 36
  Baseline (Moderate and High STEADI Risk) | 6.4 (2.7) | 6.2 (2.5)
  3 Months (All participants): number analyzed (Participants) | 58 | 48
  3 Months (All participants) | 3.3 (2.9) | 4.2 (2.8)
  3 Month (Moderate and High STEADI Risk): number analyzed (Participants) | 25 | 27
  3 Month (Moderate and High STEADI Risk) | 5.0 (3.0) | 5.2 (2.6)

6. Secondary Outcome: Modified Falls Efficacy Scale
Description: Measures fear of falling for 10 indoor and 4 outdoor activities. For each statement the participant circles a number that corresponds to their level of confidence, with zero being no confidence and 10 being extreme confidence. Once all 14 items are scored, they are added for a total score maximum of 140 which is then divided by 14. A number closer to 14 equates to more confidence, and a number closer to zero equates to less confidence.
Time Frame: 3 Months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Number analyzed (Participants) | 72 | 72
score on a scale
  Baseline (All participants): number analyzed (Participants) | 72 | 68
  Baseline (All participants) | 9.2 (1.7) | 9.0 (1.8)
  Baseline (Moderate and High STEADI Risk): number analyzed (Participants) | 43 | 35
  Baseline (Moderate and High STEADI Risk) | 8.6 (1.8) | 8.4 (2.3)
  3 Month (All participants): number analyzed (Participants) | 57 | 47
  3 Month (All participants) | 9.7 (1.1) | 9.2 (1.7)
  3 Month (Moderate and High STEADI Risk): number analyzed (Participants) | 24 | 27
  3 Month (Moderate and High STEADI Risk) | 9.6 (1.2) | 8.7 (2.1)

7. Secondary Outcome: Health Behavior Questionnaire
Description: Assessment of current behaviors related to physical activity, consuming fruits and vegetables, not smoking, and being at a recommended weight. Patients are categorized using the five levels of the trans-theoretical model of behavior change. The pre-contemplating stage, or not ready for change is scored a 5. The contemplation stage or considering making a change in the next 6 months is scored a four. The preparation or preparing to make the change in the next 6 months is scored a 3. The action stage indicates the participant has made the change and is scored. The maintenance stage indicates the participants have maintained the change for at least 6 months and are scored a 1.
Time Frame: 3 Months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Number analyzed (Participants) | 72 | 72
score on a scale
  Baseline (All participants) Physical Activity: number analyzed (Participants) | 70 | 69
  Baseline (All participants) Physical Activity | 2.0 (1.2) | 1.9 (1.3)
  Baseline (All participants) Fruit and Vegetable Consumption: number analyzed (Participants) | 71 | 66
  Baseline (All participants) Fruit and Vegetable Consumption | 2.2 (1.3) | 2.4 (1.5)
  Baseline (All participants) Smoking Habits: number analyzed (Participants) | 72 | 68
  Baseline (All participants) Smoking Habits | 1.1 (0.5) | 1.1 (.04)
  Baseline (All participants) Recommended Weight: number analyzed (Participants) | 67 | 68
  Baseline (All participants) Recommended Weight | 2.2 (1.3) | 2.2 (1.5)
  3 Month (All participants) Physical Activity: number analyzed (Participants) | 53 | 47
  3 Month (All participants) Physical Activity | 1.7 (1.0) | 2.2 (1.5)
  3 Month (All participants) Fruit and Vegetable: number analyzed (Participants) | 52 | 47
  3 Month (All participants) Fruit and Vegetable | 2.0 (1.2) | 2.2 (1.5)
  3 Month (All participants) Smoking: number analyzed (Participants) | 53 | 47
  3 Month (All participants) Smoking | 1.0 (0.3) | 1.1 (0.4)
  3 Month (All participants) Recommended Weight: number analyzed (Participants) | 52 | 46
  3 Month (All participants) Recommended Weight | 1.9 (1.2) | 1.9 (1.2)
  Baseline (Moderate and High STEADI Risk) Physical Activity: number analyzed (Participants) | 42 | 36
  Baseline (Moderate and High STEADI Risk) Physical Activity | 2.3 (1.4) | 2.3 (1.5)
  Baseline (Moderate and High STEADI Risk) Fruit and Vegetable: number analyzed (Participants) | 42 | 35
  Baseline (Moderate and High STEADI Risk) Fruit and Vegetable | 2.2 (1.3) | 2.7 (1.6)
  Baseline (Moderate and High STEADI Risk) Smoking: number analyzed (Participants) | 43 | 36
  Baseline (Moderate and High STEADI Risk) Smoking | 1.1 (0.6) | 1.1 (0.5)
  Baseline (Moderate and High STEADI Risk) Recommended Weight: number analyzed (Participants) | 40 | 36
  Baseline (Moderate and High STEADI Risk) Recommended Weight | 2.3 (1.3) | 2.5 (1.5)
  3 Month (Moderate and High STEADI Risk) Physical Activity: number analyzed (Participants) | 24 | 27
  3 Month (Moderate and High STEADI Risk) Physical Activity | 2.2 (1.2) | 2.6 (1.6)
  3 Month (Moderate and High STEADI Risk) Fruit and Vegetable: number analyzed (Participants) | 23 | 27
  3 Month (Moderate and High STEADI Risk) Fruit and Vegetable | 2.6 (1.2) | 2.3 (1.6)
  3 Month (Moderate and High STEADI Risk) Smoking: number analyzed (Participants) | 24 | 27
  3 Month (Moderate and High STEADI Risk) Smoking | 1.0 (0) | 1.0 (0)
  3 Month (Moderate and High STEADI Risk) Recommended Weight: number analyzed (Participants) | 23 | 26
  3 Month (Moderate and High STEADI Risk) Recommended Weight | 2.0 (1.4) | 2.0 (1.4)

8. Secondary Outcome: Functional Comorbidity Index
Description: Self-assessment of disease comorbidity with physical function as the outcome. 18 diagnoses are listed and if the participant has been diagnosed with the condition it would be marked at a 1 and if they do not have the condition it would be marked as a zero. Zero would be the fewest amount of co-morbidities and 18 would be the highest amount of co-morbidities.
Time Frame: 7 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Number analyzed (Participants) | 72 | 72
score on a scale
  Baseline (All participants): number analyzed (Participants) | 72 | 71
  Baseline (All participants) | 4.0 (2.1) | 3.9 (2.3)
  Baseline (Moderate and High STEADI Risk): number analyzed (Participants) | 43 | 39
  Baseline (Moderate and High STEADI Risk) | 4.7 (2.1) | 4.4 (2.4)
  3 Month (All participants): number analyzed (Participants) | 20 | 22
  3 Month (All participants) | 4.1 (2.2) | 4.5 (2.8)
  3 Month (Moderate and High STEADI Risk): number analyzed (Participants) | 7 | 13
  3 Month (Moderate and High STEADI Risk) | 5.1 (2.43) | 5.1 (3.3)
  7 Month (All participants): number analyzed (Participants) | 16 | 51
  7 Month (All participants) | 3.8 (2.6) | 4.0 (2.4)
  7 Month (Moderate and High STEADI Risk): number analyzed (Participants) | 3 | 23
  7 Month (Moderate and High STEADI Risk) | 5.0 (1.0) | 4.6 (2.8)

9. Secondary Outcome: Home Falls and Accidents Screening Tool (Home FAST)
Description: The tool evaluates 25 home safety domains and includes questions related to lighting, floor surfaces, and properly fitted foot wear. The original tool design was not scored but the investigators have added a scoring system (13 = safest environment to 50 = least safe environment) to quantify each question pertaining to the home environment. 13 home safety questions are scored as either Yes (indicating the recommended safety modifications was present) or No (indicating the recommended safety modifications had not been met). An additional 12 questions have an N/A option to be used in circumstances where a condition was not met (e.g., participant does not have a pet or stairs in the home). The investigators coded the responses as YES=1 point, NO= 2 points, an N/A= null within that category and not included during calculation. Therefore, overall Home FAST scores that decrease over time would suggest diminished home fall and accident risks related to their environment.
Time Frame: 7 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Number analyzed (Participants) | 72 | 72
score on a scale
  Baseline (All participants): number analyzed (Participants) | 70 | 69
  Baseline (All participants) | 25.7 (6.2) | 25.9 (7.8)
  Baseline (Moderate and High STEADI Risk): number analyzed (Participants) | 42 | 39
  Baseline (Moderate and High STEADI Risk) | 25.5 (6.7) | 24.9 (8.6)
  3 Month (All participants): number analyzed (Participants) | 54 | 45
  3 Month (All participants) | 25.6 (5.7) | 26.8 (7.3)
  3 Month (Moderate and High STEADI Risk): number analyzed (Participants) | 25 | 27
  3 Month (Moderate and High STEADI Risk) | 25.4 (6.2) | 26.3 (8.5)
  7 Month (All participants): number analyzed (Participants) | 47 | 41
  7 Month (All participants) | 26.0 (5.0) | 25.6 (5.9)
  7 Month (Moderate and High STEADI Risk): number analyzed (Participants) | 16 | 19
  7 Month (Moderate and High STEADI Risk) | 26.9 (5.7) | 23.4 (5.5)

10. Secondary Outcome: Body Mass Index
Description: Assessment of body fat calculated from height and weight.
Time Frame: 7 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Number analyzed (Participants) | 72 | 72
kg/m^2
  Baseline (All participants): number analyzed (Participants) | 72 | 68
  Baseline (All participants) | 29.9 (5.4) | 28.6 (5.4)
  Baseline (Moderate and High STEADI Risk): number analyzed (Participants) | 43 | 37
  Baseline (Moderate and High STEADI Risk) | 30.2 (5.4) | 29.2 (5.6)
  7 Month (All participants): number analyzed (Participants) | 11 | 47
  7 Month (All participants) | 29.5 (5.2) | 35.1 (4.1)
  7 Month (Moderate and High STEADI Risk): number analyzed (Participants) | 24 | 20
  7 Month (Moderate and High STEADI Risk) | 32.7 (1.1) | 30.9 (6.0)

11. Secondary Outcome: Blood Pressure
Description: Assessment of mean resting blood pressure in seated position.
Time Frame: 7 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Number analyzed (Participants) | 72 | 72
mm Hg
  Baseline (All participants) Systolic: number analyzed (Participants) | 72 | 71
  Baseline (All participants) Systolic | 133 (20) | 131 (15)
  Baseline (All participants) Diastolic: number analyzed (Participants) | 72 | 71
  Baseline (All participants) Diastolic | 76 (10) | 78 (10)
  Baseline (Moderate and High STEADI Risk) Systolic: number analyzed (Participants) | 43 | 39
  Baseline (Moderate and High STEADI Risk) Systolic | 133 (22) | 132 (15)
  Baseline (Moderate and High STEADI Risk) Diastolic: number analyzed (Participants) | 43 | 39
  Baseline (Moderate and High STEADI Risk) Diastolic | 76 (10) | 79 (12)
  3 Month (All participants) Systolic: number analyzed (Participants) | 64 | 58
  3 Month (All participants) Systolic | 125 (15) | 125 (22)
  3 Month (All participants) Diastolic: number analyzed (Participants) | 64 | 58
  3 Month (All participants) Diastolic | 76 (15) | 75 (10)
  3 Month (Moderate and High STEADI Risk) Systolic: number analyzed (Participants) | 29 | 32
  3 Month (Moderate and High STEADI Risk) Systolic | 123 (13) | 123 (21)
  3 Month (Moderate and High STEADI Risk) Diastolic: number analyzed (Participants) | 29 | 32
  3 Month (Moderate and High STEADI Risk) Diastolic | 74 (8) | 74 (7)
  7 Month (All participants) Systolic: number analyzed (Participants) | 54 | 51
  7 Month (All participants) Systolic | 128 (19) | 128 (16)
  7 Month (All participants) Diastolic: number analyzed (Participants) | 54 | 51
  7 Month (All participants) Diastolic | 76 (10) | 75 (10)
  7 Month (Moderate and High STEADI Risk) Systolic: number analyzed (Participants) | 16 | 23
  7 Month (Moderate and High STEADI Risk) Systolic | 127 (18) | 126 (16)
  7 Month (Moderate and High STEADI Risk) Diastolic: number analyzed (Participants) | 16 | 23
  7 Month (Moderate and High STEADI Risk) Diastolic | 75 (10) | 75 (11)

12. Secondary Outcome: Number of Participants With Orthostatic Hypotension
Description: Blood pressure was measured sequentially in supine, seated and standing and orthostatic hypotension was determined by the following parameters: a systolic blood pressure decrease of greater than or equal to 20 mm Hg or a diastolic blood pressure decrease of greater than or equal to 10 mm Hg between any of the three positions after three minutes in that position.
Time Frame: 7 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
Number analyzed (Participants) | 72 | 72
Participants
  Baseline (All participants): number analyzed (Participants) | 72 | 71
  Baseline (All participants) | 13 | 16
  Baseline (Moderate and High Fall Risk Participants): number analyzed (Participants) | 43 | 39
  Baseline (Moderate and High Fall Risk Participants) | 10 | 12
  3 Month (All Participants: number analyzed (Participants) | 62 | 58
  3 Month (All Participants | 13 | 7
  3 Month (Moderate and High Fall Risk Participants): number analyzed (Participants) | 28 | 32
  3 Month (Moderate and High Fall Risk Participants) | 4 | 3
  7 Month (All Participants): number analyzed (Participants) | 53 | 51
  7 Month (All Participants) | 10 | 5
  7 Month (Moderate and High Fall Risk Participants): number analyzed (Participants) | 15 | 23
  7 Month (Moderate and High Fall Risk Participants) | 4 | 2

ADVERSE EVENTS:
Time Frame: 1 year 4 months
Description: The most likely adverse event for this population would be falls.
Arm/Group | HOP-UP-PT Program | Normal Level of Activity
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 0/72 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT04814459/Prot_SAP_001.pdf